CLINICAL TRIAL: NCT06001840
Title: Promotion and Mitigation Factors Leading to Illegal Tobacco Purchases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 5P01CA200512 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking; Nicotine Vaping
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: We will examine two promotion policies. In the full nicotine conditions, participants' preferred cigarettes and NVP products will be available in the LETM and preferred cigarettes will be available in the iETM. In the low nicotine conditions, a ban will permit only very-low nicotine cigarettes (VLNCs) in the LETM and preferred cigarettes will be available in the iETM. Additionally, we will model three mitigation strategies that may reduce iETM purchases: health communications, availability of nicotine replacement, and penalties. The three mitigation factors will be applied during both promotion policies described above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Exclusive cigarette smokers (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Behavioral: Promotion factors; Behavioral: Mitigation strategies
- Experimental: Dual cigarette/ nicotine vaping product users (Experimental): Dual cigarette and nicotine vaping product users will be recruited and will be exposed to all of the conditions described in the intervention section
  Interventions: Behavioral: Promotion factors; Behavioral: Mitigation strategies

INTERVENTIONS:
Behavioral: Promotion factors — In the full nicotine conditions, participants' preferred cigarettes and NVP products will be available in the LETM and preferred cigarettes will be available in the iETM. In the low nicotine conditions, a ban will permit only VLNCs in the LETM and preferred cigarettes will be available in the iETM.
Behavioral: Mitigation strategies — Penalties: Penalties will be presented as a 60% chance of getting caught making illegal purchases. The consequences of illegal purchases include not receiving any study products from the ETM if they were caught and randomly drew that trial.

SUMMARY:
This study will investigate the effects of promotion factors and mitigation strategies on legal and illegal tobacco purchases for different tobacco-user types.

DETAILED DESCRIPTION:
In the present study, we propose to examine some promotion factors and mitigation strategies and how they impact tobacco product legal and illegal purchases. Specifically, we have developed an Illegal Experimental Tobacco Marketplace (iETM). The iETM permits us to identify the number, type, and characteristics of tobacco users who would seek illegal tobacco products and the conditions that would induce them to seek that option. The critical questions we seek to answer are whether changes in product standards and availability will engender illegal tobacco purchasing as a function of tobacco user type (e.g., exclusive combustible product users, and dual cigarette/NVP users). Understanding the user types and the relevant conditions will inform greater tailoring of policy to diminish consumer interest in an illegal market.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Be at least 21 years of age or older
* Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm)
* Stable tobacco use patterns for at least two months

For exclusive cigarette smokers:

* Smoke at least 10 cigarettes daily and do not use NVPs regularly (no more than 9 times in the last month).
* For dual cigarette/NVP users:
* Smoke at least 10 cigarettes daily and use NVPs at least 3 times in a week (report use of closed nicotine salt system)

Exclusion criteria:

* Have plans to move out of the area
* Have a serious or unstable physical or mental health condition
* Taking a tobacco cessation medication or medication that interferes with nicotine metabolism, motivation or reinforcement
* Report concrete, immediate plans to alter/quit using their usual nicotine products at the beginning of the study
* Being pregnant or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas-Lemos, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at Virginia Tech Carilion
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Exclusive Cigarette Smokers; Experimental: Dual Cigarette/ Nicotine Vaping Product Users: Participants completed four within-subject ETM conditions (No Policy; Penalty Only; VLNC Only; Penalty + VLNC) in a randomized, counterbalanced order.
Period: Overall Study
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Started | 33 | 32
No Policy | 27 | 26
Penalty Only | 31 | 29
VLNC Only | 27 | 26
Penalty + VLNC | 31 | 29
Completed | 27 | 26
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Screen fail | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Exclusive Cigarette Smokers: Exclusive Cigarette Smokers completed all four within-subject experimental conditions described in the intervention section, presented in a randomized, counterbalanced order. Within each condition, participants completed five trials in which the market price of legal cigarettes systematically increased from ½×, 1×, 2×, 4×, to 8× , allowing evaluation of purchasing behavior under escalating prices. Sequences of conditions were not tracked. Milestones (conditions) are used to indicate exposure without double-counting participants.
  Promotion Factors:
  In full nicotine conditions, participants' preferred cigarettes were available in the Legal Experimental Tobacco Marketplace (LETM), while preferred cigarettes were also available in the Illegal Experimental Tobacco Marketplace (iETM).
  In low nicotine conditions, very low nicotine content (VLNC) cigarettes were available in the LETM, while preferred cigarettes remained available in the iETM.
  Mitigation Strategy:
  Penalties simulated enforcement with a 60% likelihood of being "caught" making an illegal purchase. If caught, participants left the session without products.
  No Policy: Full nicotine cigarettes available in LETM; no penalty.
  Penalty Only: Full nicotine cigarettes available in LETM; 60% chance of being caught.
  VLNC Only: Only VLNC cigarettes available in LETM; no penalty.
  Penalty + VLNC: VLNC cigarettes only in LETM; 60% chance of being caught.
- Experimental: Dual Cigarette/ Nicotine Vaping Product Users: Duak completed all four within-subject experimental conditions described in the intervention section, presented in a randomized, counterbalanced order. Within each condition, participants completed five trials in which the market price of legal cigarettes systematically increased from ½×, 1×, 2×, 4×, to 8× , allowing evaluation of purchasing behavior under escalating prices. Sequences of conditions were not tracked. Milestones (conditions) are used to indicate exposure without double-counting participants.
  Promotion Factors:
  In full nicotine conditions, participants' preferred cigarettes were available in the Legal Experimental Tobacco Marketplace (LETM), while preferred cigarettes were also available in the Illegal Experimental Tobacco Marketplace (iETM).
  In low nicotine conditions, very low nicotine content (VLNC) cigarettes were available in the LETM, while preferred cigarettes remained available in the iETM.
  Mitigation Strategy:
  Penalties simulated enforcement with a 60% likelihood of being "caught" making an illegal purchase. If caught, participants left the session without products.
  No Policy: Full nicotine cigarettes available in LETM; no penalty.
  Penalty Only: Full nicotine cigarettes available in LETM; 60% chance of being caught.
  VLNC Only: Only VLNC cigarettes available in LETM; no penalty.
  Penalty + VLNC: VLNC cigarettes only in LETM; 60% chance of being caught.
- Total: Total of all reporting groups
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.74 (9.02) | 43.15 (8.04) | 43.94 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 18 | 18 | 36
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Household Income [Count of Participants; unit: Participants]
  Less than $19,000 | 18 | 18 | 36
  $20,000-$39,999 | 4 | 5 | 9
  $40,000-$64,999 | 1 | 3 | 4
  $65,000-$99,999 | 2 | 0 | 2
  $100,000-$154,999 | 2 | 0 | 2
  Greater than $155,000 | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  < 12 years | 4 | 2 | 6
  12 years | 8 | 8 | 16
  13-15 years | 12 | 13 | 25
  16+ years | 3 | 3 | 6
Timeline Follow Back (TLFB)- Cigarettes [Mean (Standard Deviation); unit: cigarettes per day] — The Timeline Followback is an assessment tool to measure tobacco use. This is formatted as a calendar, where individuals retrospectively estimate their past 30-day tobacco/nicotine use. They report the amount consumed each day (e.g., number of cigarettes, ) during the past 30 days. These are then averaged to get a mean and SD.
  cigarettes per day | 19.95 (7.77) | 17.71 (0.76) | 18.83 (4.26)
ETM Budget [Mean (Standard Deviation); unit: dollars per week] — The ETM budget is calculated to estimate weekly expenditure. This is based on the average values from the timeline follow-back for the past 30-day tobacco/nicotine use. The average is then multiplied by the cost of the product and then multiplied by 7 to get a weekly budget. This is then used in the Experimental Tobacco Marketplace (ETM) as the amount of money they can use to purchase products.
  dollars per week | 53.10 (25.0) | 71.5 (28.2) | 62.3 (26.6)
Heaviness of Smoking Index (HSI) [Mean (Standard Deviation); unit: units on a scale] — The Heaviness of Smoking Index (HSI) was developed as a test to measure nicotine dependence by using two questions: time to first smoking in the morning and number of cigarettes per day. It uses a six-point scale calculated from the number of cigarettes smoked per day (1-10, 11-20, 21-30, 31+) and the time to first cigarette after waking (less than/equal to 5, 6-30, 31-60, and 61+ minutes). Nicotine dependence is then categorized into a three-category variable: low (0-1), medium (2-4), and high (5-6).
  units on a scale | 4.04 (1.09) | 3.81 (2.56) | 3.93 (1.83)
Questionairre on Smoking Urges (QSU)- brief [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The Questionnaire of Smoking Urges - Brief (QSU-Brief) is a 10-item measure used to assess craving to smoke. Participants rate each statement on a 7-point Likert scale, ranging from "strongly disagree" (1) to "strongly agree" (7). Total scores range from 10 to 70, with higher scores indicating a stronger urge to smoke. We summed each participant's responses to obtain total scores, then calculated the group mean and standard deviation.
  units on a scale
    Cigarettes | 47.93 (15.77) | 50.42 (13.96) | 49.18 (14.87)
    E-cigarettes | 17.22 (12.58) | 41.81 (15.19) | 29.52 (13.89)
Intention to quit cigarettes [Mean (Standard Deviation); unit: units on a scale] — Intention to quit is a one-item questionnaire with a slider (scale 0-10). 0=no thought of quitting, 5=thinking about quitting but not quite ready, and 10=taking action to quit (e.g., setting quit date). Higher score represent higher intention to quit.
  units on a scale | 6.50 (2.43) | 6.00 (1.41) | 6.25 (1.92)
Timeline Follow Back (TLFB)- E-cigarettes [Mean (Standard Deviation); unit: mL per day] — The Timeline Followback is an assessment tool to measure tobacco use. This is formatted as a calendar, where individuals retrospectively estimate their past 30-day tobacco/nicotine use. They report the amount consumed each day (e.g., mL per day,. # of puffs, ) during the past 30 days. These are then averaged to get a mean and SD.
  mL per day | 0.00 (0.01) | 0.98 (1.42) | 0.49 (0.72)
Heavines of Vaping Index (HVI) [Mean (Standard Deviation); unit: units on a scale] — The Heaviness of Vaping Index (HVI) was developed as a test to measure nicotine dependence by using two questions: time to first smoking in the morning and number of cigarettes per day. It uses a six-point scale calculated from the number of cigarettes smoked per day (1-10, 11-20, 21-30, 31+) and the time to first cigarette after waking (less than/equal to 5, 6-30, 31-60, and 61+ minutes). Nicotine dependence is then categorized into a three-category variable: low (0-1), medium (2-4), and high (5-6). Population: We did not collect this measure from exclusove cigarette users as they previously reported no e-cigarette use.
  units on a scale
    number analyzed (Participants) | 0 | 26 | 26
    (all) |  | 2.56 (2.29) | 2.56 (2.29)
Intention to quit e-cigarettes [Mean (Standard Deviation); unit: units on a scale] — Intention to quit is a one-item questionnaire with a slider (scale 0-10). 0=no thought of quitting, 5=thinking about quitting but not quite ready, and 10=taking action to quit (e.g., setting quit date). Higher score represent higher intention to quit. Population: We did not collect this measure for exclusive cigarette users as they preveiously reported no e-cigarette use.
  units on a scale
    number analyzed (Participants) | 0 | 26 | 26
    (all) |  | 2.24 (2.54) | 2.24 (2.54)

OUTCOME MEASURES:

1. Primary Outcome: Percent Budget Spent on Illegal Cigarettes Across Policy Conditions
Description: The study has 4 policy conditions with combinations of promotion strategy (VLNC standard) and mitigation strategy (penalties), and each combination: No Policy, Penalty only, VLNC only, and Penalty + VLNC. The average percentage of the budget spent on illegal cigarettes across all trials was calculated for each policy scenario.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of budget spent
Groups:
- Experimental: Dual Cigarette/ Nicotine Vaping Product Users: Dual users completed all four within-subject experimental conditions described in the intervention section, presented in a randomized, counterbalanced order. Within each condition, participants completed five trials in which the market price of legal cigarettes systematically increased from ½×, 1×, 2×, 4×, to 8× , allowing evaluation of purchasing behavior under escalating prices. Sequences of conditions were not tracked. Milestones (conditions) are used to indicate exposure without double-counting participants.
  Promotion Factors:
  In full nicotine conditions, participants' preferred cigarettes were available in the Legal Experimental Tobacco Marketplace (LETM), while preferred cigarettes were also available in the Illegal Experimental Tobacco Marketplace (iETM).
  In low nicotine conditions, very low nicotine content (VLNC) cigarettes were available in the LETM, while preferred cigarettes remained available in the iETM.
  Mitigation Strategy:
  Penalties simulated enforcement with a 60% likelihood of being "caught" making an illegal purchase. If caught, participants left the session without products.
  No Policy: Full nicotine cigarettes available in LETM; no penalty.
  Penalty Only: Full nicotine cigarettes available in LETM; 60% chance of being caught.
  VLNC Only: Only VLNC cigarettes available in LETM; no penalty.
  Penalty + VLNC: VLNC cigarettes only in LETM; 60% chance of being caught.
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 27 | 26
percentage of budget spent
  No Policy | 40.78 (4.04) | 38.41 (3.63)
  Penalty only | 12.14 (2.66) | 9.64 (2.32)
  VLNC only | 71.20 (3.42) | 65.18 (2.84)
  Penalty + VLNC | 26.31 (3.47) | 20.94 (3.09)

2. Primary Outcome: Percent Budget Spent on Legal Cigarettes Across Policy Conditions
Description: The study has 4 policy conditions with combinations of promotion strategy (VLNC standard) and mitigation strategy (penalties), and each combination: No Policy, Penalty only, VLNC only, and Penalty + VLNC. The average percentage of the budget spent on legal cigarettes across all trials was calculated for each policy scenario.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of budget spent
Groups:
- Experimental: Exclusive Cigarette Smokers: Exclusive Cigarette Smokers (no regular vape product use) completed all four within-subject experimental conditions described in the intervention section, presented in a randomized, counterbalanced order. Within each condition, participants completed five trials in which the market price of legal cigarettes systematically increased from ½×, 1×, 2×, 4×, to 8× , allowing evaluation of purchasing behavior under escalating prices. Sequences of conditions were not tracked. Milestones (conditions) are used to indicate exposure without double-counting participants.
  Promotion Factors:
  In full nicotine conditions, participants' preferred cigarettes were available in the Legal Experimental Tobacco Marketplace (LETM), while preferred cigarettes were also available in the Illegal Experimental Tobacco Marketplace (iETM).
  In low nicotine conditions, very low nicotine content (VLNC) cigarettes were available in the LETM, while preferred cigarettes remained available in the iETM.
  Mitigation Strategy:
  Penalties simulated enforcement with a 60% likelihood of being "caught" making an illegal purchase. If caught, participants left the session without products.
  No Policy: Full nicotine cigarettes available in LETM; no penalty.
  Penalty Only: Full nicotine cigarettes available in LETM; 60% chance of being caught.
  VLNC Only: Only VLNC cigarettes available in LETM; no penalty.
  Penalty + VLNC: VLNC cigarettes only in LETM; 60% chance of being caught.
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 27 | 26
percentage of budget spent
  No Policy | 37.97 (3.73) | 29.72 (3.28)
  Penalty only | 57.30 (3.59) | 47.73 (3.30)
  VLNC only | 4.32 (1.31) | 0.89 (0.37)
  Penalty + VLNC | 19.71 (2.84) | 9.69 (2.06)

3. Primary Outcome: Percent Budget Spent on E-cigarettes Across Policy Conditions
Description: The study has 4 policy conditions with combinations of promotion strategy (VLNC standard) and mitigation strategy (penalties), and each combination: No Policy, Penalty only, VLNC only, and Penalty + VLNC. The average percentage of the budget spent on e-cigarettes across all trials was calculated for each policy scenario.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of budget spent
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 27 | 26
percentage of budget spent
  No Policy | 10.01 (1.48) | 23.06 (2.27)
  Penalty only | 20.16 (2.56) | 27.15 (2.41)
  VLNC only | 11.49 (1.71) | 24.06 (2.39)
  Penalty + VLNC | 37.63 (3.12) | 46.51 (3.16)

4. Primary Outcome: Percent Budget Spent on Nicotine Replacement Therapy Across Policy Conditions
Description: The study has 4 policy conditions with combinations of promotion strategy (VLNC standard) and mitigation strategy (penalties), and each combination: No Policy, Penalty only, VLNC only, and Penalty + VLNC. The average percentage of the budget spent on nicotine replacement theray across all trials was calculated for each policy scenario.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of budget spent
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 27 | 26
percentage of budget spent
  No Policy | 2.00 (0.44) | 3.67 (0.86)
  Penalty only | 3.11 (0.70) | 4.56 (0.91)
  VLNC only | 3.46 (0.94) | 4.38 (1.10)
  Penalty + VLNC | 8.71 (1.41) | 6.89 (1.08)

5. Primary Outcome: Percent Budget Spent on Oral Nicotine/Tobacco Across Policy Conditions
Description: The study has 4 policy conditions with combinations of promotion strategy (VLNC standard) and mitigation strategy (penalties), and each combination: No Policy, Penalty only, VLNC only, and Penalty + VLNC. The average percentage of the budget spent on oral nicotine/tobacco across all trials was calculated for each policy scenario.
Time Frame: 1 day
Measure: Mean (Standard Error); unit: percentage of budget spent
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 27 | 26
percentage of budget spent
  No Policy | 0.85 (0.40) | 0.12 (0.05)
  Penalty only | 0.69 (0.32) | 0.89 (0.63)
  VLNC only | 1.08 (0.50) | 0.21 (0.09)
  Penalty + VLNC | 0.71 (0.31) | 0.37 (0.11)

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Experimental: Exclusive Cigarette Smokers: Exclusive cigarette smokers will be recruited and will be exposed to all of the conditions described in the intervention section.
  Promotion factors: In the full nicotine conditions, participants' preferred cigarettes and NVP products will be available in the LETM and preferred cigarettes will be available in the iETM. In the low nicotine conditions, a ban will permit only VLNCs in the LETM and preferred cigarettes will be available in the iETM.
  Mitigation strategies: Health Communications. The first narrative describes a person unknown to the participant who purchases from the illegal market and experiences negative life outcomes (e.g., ill health from contaminants). The second narrative incorporates cognitive biases of social proof (i.e., portraying a choice as the opinion of the majority).
  Availability of Nicotine Replacement Therapies (NRT): Transdermal NRT will be available in the LETM at two different prices. In one condition, transdermal NRT will be available at a 50% subsidy in the form of coupons. In the other condition, a five-day supply of NRT will be available for free.
  Penalties: Penalties will be presented in different fine magnitudes along with a description of the consequences of illegal purchases (i.e., a criminal record).
- Experimental: Dual Cigarette/ Nicotine Vaping Product Users: Dual cigarette and nicotine vaping product users will be recruited and will be exposed to all of the conditions described in the intervention section
  Promotion factors: In the full nicotine conditions, participants' preferred cigarettes and NVP products will be available in the LETM and preferred cigarettes will be available in the iETM. In the low nicotine conditions, a ban will permit only VLNCs in the LETM and preferred cigarettes will be available in the iETM.
  Mitigation strategies: Health Communications. The first narrative describes a person unknown to the participant who purchases from the illegal market and experiences negative life outcomes (e.g., ill health from contaminants). The second narrative incorporates cognitive biases of social proof (i.e., portraying a choice as the opinion of the majority).
  Availability of Nicotine Replacement Therapies (NRT): Transdermal NRT will be available in the LETM at two different prices. In one condition, transdermal NRT will be available at a 50% subsidy in the form of coupons. In the other condition, a five-day supply of NRT will be available for free.
  Penalties: Penalties will be presented in different fine magnitudes along with a description of the consequences of illegal purchases (i.e., a criminal record).
Arm/Group | Experimental: Exclusive Cigarette Smokers | Experimental: Dual Cigarette/ Nicotine Vaping Product Users
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT06001840/Prot_SAP_ICF_000.pdf